CLINICAL TRIAL: NCT02906956
Title: Music and Adherence in Upper Extremity Home Programs Post Stroke
Brief Title: Music and Adherence Home Programs Post Stroke
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2016/06/18
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preferred Music Playlist (Experimental): All participants will have this phase twice in the protocol. See description in intervention section.
  Interventions: Behavioral: Preferred music playlist

INTERVENTIONS:
Behavioral: Preferred music playlist — Client will be instructed in a home program based on repetitive task practice principles and will complete this program with and without the use of a preferred music playlist during practice.

SUMMARY:
The purpose of this study is to explore whether adherence to upper extremity home programs changes when persons post stroke practice with preferred music.

ELIGIBILITY:
Inclusion Criteria:

* Ages 40-85
* Mild to Moderate hemiparesis as determined by a score of 21 to 50 on the FM- UE
* At least 6 months post stroke
* American English as primary language

Exclusion Criteria:

* Significant visual impairment as determined by "aphasia-friendly" and age appropriate screening
* Significant hearing impairment as determined by self-report
* Actively receiving occupational or physical therapy services for upper extremity motor recovery
* Severe auditory comprehension impairment such that they cannot understand one-step directions as indicated by a WAB-R score below 8/10 on Sequential Commands Subtest
* Sitting or standing blood pressure of 180/110 or HE > 100 bpm

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of sessions of practice | 4 weeks
Duration of sessions of practice | 4 weeks
Number of minutes of practice | 4 weeks

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline and no more than one week post intervention period
  Perceived occupational performance on activities of importance to the client
Motor Activity Log | Baseline and no more than one week post intervention period
  Perceived amount and quality of use of the affected upper extremity
Western Aphasia Battery - Revised | Baseline
  Measure of language impairment
Cognitive Linguistic Quick Test | Baseline
  Measure of cognition

OTHER OUTCOMES:
Qualitative Feedback Interview | No more than 3 weeks post intervention period
  One-to-one interview with supported communication strategies on the experience of the intervention and study materials.
Intensity of Practice | 4 weeks
  Rate of accelerations as measured by an activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Elena V Donoso Brown, PhD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University Speech, Hearing, Language Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No